CLINICAL TRIAL: NCT00794482
Title: A Multi-centre, Multi-national Open Study in Patients With Hepatic Cirrhosis to Characterise the Association Between the Pharmacokinetics of NRL972 and Disease Severity.
Brief Title: Multi-national Cirrhosis Study to Characterise the Association Between the Pharmacokinetics of NRL972 and Disease Severity.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Vice President, Clinical Development, Norgine Ltd
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NRL972-03/2006 (CIR)
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2009-10

CONDITIONS: Hepatic Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — NRL972

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: NRL972 — Single dose of 2 mg NRL972 administered intravenously. Total volume 5 mL.

SUMMARY:
This is a multi-centre, multi-national, open study to assess the pharmacokinetics of NRL972 in patients with hepatic cirrhosis CTP-classes A, B, and C (histologically confirmed by liver biopsy). The pharmacokinetics of NRL972 will be referenced to a Clinical Staging Matrix obtained during a clinical work-up of patients with hepatic cirrhosis. Patients to be studied will have histologically established hepatic cirrhosis or confirmed hepatic cirrhosis by an objective imaging study without confounding end-stage co-morbidity. Within 14 days of confirming eligibility, the investigations will be conducted over 2-5 days with the test procedures (clinical laboratory tests, ultrasound (US)-investigations, gastroscopy, NRL972- and MEGX'-test). Up to one week after the NRL972-test, a follow-up telephone call will be made.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting the following conditions will be eligible for enrolment:

* Patient has given his or her written informed consent to the study participation, prior to study specific procedures
* Male and female (non-child-bearing potential = post-menopausal or medically adequate contraception)
* Ethnicity: any
* Age: 18 to 80 years of age
* Patients with histologically established diagnosis of hepatic cirrhosis and available histological material for review by the central histopathologist or a CTP score greater than or equal to 10 points plus an objective imaging study (CT or NMR scan) within 3 months of the screening visit with a confirmation of hepatic cirrhosis (scans are collected and reviewed), but excluding patients with the diagnosis of primary biliary cirrhosis, primary sclerosing cholangitis and cystic fibrosis-associated liver disease
* Present CTP-class A, B or C
* Medically fit to undergo the protocol-defined procedures without undue risk and discomfort
* Predicted life-expectancy greater than or equal to 6 months by clinical judgement

Exclusion Criteria:

Subjects of any of the following categories will be excluded from enrolment:

* Previous participation in this trial (except for scheduled re-testing in relation to technical difficulties with initial test)
* Participant in any other trial during the last 90 days
* Donation of blood during the last 60 days or a history of blood loss exceeding 300 mL within the last 3 months
* Any donation of germ cells, blood, organs, or bone marrow during the course of the study
* History of any clinically relevant allergy (including hypersensitivity to the trial medications)
* Presence of clinical relevant acute or chronic infection (other than chronic viral hepatitis, if applicable)
* Use of confounding concomitant medication
* Presence or history of any end-stage (co-)morbidity (excluding the effects of hepatic cirrhosis) such as: malignancy and clinically relevant systemic diseases
* Suspicion or evidence that the subject is not trustworthy and reliable
* Suspicion or evidence that the subject is not able to make a free consent or to understand the information in this regard
* Primary biliary cirrhosis and primary sclerosing cholangitis
* Cystic fibrosis
* Previous liver transplantation or intended liver transplantation within 6 months after enrolment
* Patients having undergone previous transjugular intrahepatic portosystemic shunt (TIPS) or portocaval anastomosis (PCA)
* Patients who are employees at the investigational site, relatives or spouses of the investigator
* Current drug, or medication abuse

Special restrictions for female patients:

* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means, unless they meet the following definition of post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels greater than 40 mIU/m or 6 weeks post surgical bilateral oophorectomy with or without hysterectomy or hysterectomy or are using one or more of the following acceptable methods of contraception: surgical sterilization (e.g., bilateral tubal ligation, vasectomy), hormonal contraception (implantable, patch, oral), and double-barrier methods (any double combination of: IUD, male or female condom with spermicidal gel, diaphragm, sponge, cervical cap)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Influence of CTP staging on the pharmacokinetics of NRL972 in patients with cirrhosis. | Single dose, 2-5 day follow-up

SECONDARY OUTCOMES:
Inter-subject relationship between the pharmacokinetics of NRL972 and other parameters used to define the severity of hepatic cirrhosis | 2-5 days
To assess the safety and tolerability of 2mg NRL972 administered by intravenous injection to patients with hepatic cirrhosis | 2-5 days

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Essen, Germany